CLINICAL TRIAL: NCT04278170
Title: An Investigation of Factors Affecting Sleep Quality in Patients With Rheumatoid Arthritis
Brief Title: Sleep Quality in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: TURKEYPMRTRH
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Rheumatoid Arthritis
Keywords: sleeping disorders; sleep quality
MeSH Terms: conditions — Arthritis, Rheumatoid; Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case group: Rheumatoid arthritis patients who met the American College of Rheumatology (ACR) 2010 RA classification
  Interventions: Other: no attempt was made to patients

INTERVENTIONS:
Other: no attempt was made to patients — no attempt was made to patients

SUMMARY:
This study was designed to investigate the factors affecting sleep quality of Rheumatoid arthritis patients in Turkish population.

DETAILED DESCRIPTION:
Demographic data, duration of disease, routine biochemical tests and currently used medications were recorded. Disease activity was assessed with Disease Activity Score 28 (DAS 28). Visual Analog Scale (VAS) was used to evaluate pain levels. Health Assessment Questionnaire (HAQ) was used to assess activities of daily living. Beck depression inventory (BDI) was used to investigate the signs of depression in patients. Sleep quality was considered to be poor in patients with a Pittsburgh Sleep Quality Index (PSQI) global score of 5 and greater.

ELIGIBILITY:
Inclusion Criteria:

* patients with RA who met the 2010 American College of Rheumatology (ACR) RA classification criteria were included

Exclusion Criteria:

* Patients who had difficulties understanding and responding to questions were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
The factor affecting sleep quality of Rheumatoid arthritis patients | 1 day
  Demographic data
duration of disease | 1 day
  factor affecting sleep quality of Rheumatoid arthritis patients
Sleep quality of Rheumatoid arthritis patients | 1 day
  Pittsburg Sleep Quality Index (PSQI) was used to evaluate the sleep quality of the patients. PSQI is a questionnaire which assesses sleep quality by questioning the patient on 7 main sections; i.e., subjective sleep quality, sleep latency, sleep duration, habitual sleep activity, sleep disorders, use of sleep medication and daytime dysfunctions. Questions are scored from 0 to 3, high scores reflecting poor sleep quality. Seven main components are first evaluated individually and then the scores are added. A total score of 5 and above indicates poor sleep quality
Disease activity of Rheumatoid arthritis patients | 1 day
  Disease activity was assessed with Disease Activity Score 28 (DAS 28).
The pain evaluating of Rheumatoid arthritis patients | 1 day
  Visual Analog Scale (VAS) was used to evaluate pain levels.
General health of Rheumatoid arthritis patients | 1 day
  Health Assessment Questionnaire (HAQ) was used to assess activities of daily living.
Depression of Rheumatoid arthritis patients | 1 day
  Beck depression inventory (BDI) was used to investigate the signs of depression in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Bardak, MD, Study Director — Istanbul Physical Therapy and Rehabilitation Research and Training Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Szady P, Baczyk G, Kozlowska K. Fatigue and sleep quality in rheumatoid arthritis patients during hospital admission. Reumatologia. 2017;55(2):65-72. doi: 10.5114/reum.2017.67600. Epub 2017 Apr 28. PMID 28539677
- [Background] Purabdollah M, Lakdizaji S, Rahmani A, Hajalilu M, Ansarin K. Relationship between Sleep Disorders, Pain and Quality of Life in Patients with Rheumatoid Arthritis. J Caring Sci. 2015 Sep 1;4(3):233-41. doi: 10.15171/jcs.2015.024. eCollection 2015. PMID 26464840
- [Background] Goes ACJ, Reis LAB, Silva MBG, Kahlow BS, Skare TL. Rheumatoid arthritis and sleep quality. Rev Bras Reumatol Engl Ed. 2017 Jul-Aug;57(4):294-298. doi: 10.1016/j.rbre.2016.07.011. Epub 2016 Aug 12. English, Portuguese. PMID 28743355